CLINICAL TRIAL: NCT02621268
Title: A Pilot & Feasibility Study of the Imaging Potential of Indocyanine Green in Subjects Undergoing Minimally Invasive Thoracic Surgery Presenting With Thoracic Nodules
Brief Title: Minimally Invasive Imagery With Indocyanine Green
Acronym: ICG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sunil Singhall, Director, Thoracic Surgery Research Laboratory, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 820766
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indocyanine Green (Experimental): Dosage calculated by weight of individual, 5mg/kg.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Infusion of ICG 24 hours prior to surgery
  Other Names: ICG

SUMMARY:
Determine if ICG administered pre-operatively, then imaged intraoperatively using our cameras, will aid in the identification of a suspected thoracic nodules, margins, lymph nodes and satellite nodules during minimally invasive procedures. The investigators intend on enrolling 48 Subjects in this study. The study is focusing on patients presenting with suspected thoracic cancers who are considered to be good minimally invasive surgical candidates

DETAILED DESCRIPTION:
According to the World Health Organization, lung cancer is the most common cause of cancer-related death in men and women, and is responsible for 1.3 million deaths worldwide annually as of 2004.

Surgery remains the best option for patients presenting with operable Stage I or II cancers, however the five year survival rate for these candidates remains at a dismal 53% for Stage I and 32% for Stage II (1). The high rates of recurrence suggest that surgeons are unable to completely detect and remove primary tumor nodules in a satisfactory manner as well as lingering metastases in sentinel lymph nodes. By ensuring a negative margin through near-infrared imagery it would be possible for us to improve the rates of recurrence free patients and thus overall survival.

The use of an ICG probe will allow for the operating field and lung tissue to be observed in real-time.

ICG has been used in the clinical settings since 1957. There is a wealth of data available attesting to the safety of this drug injected at its current clinically indicated dosing level. ICG has been shown to preferentially uptake in esophageal tumors as opposed to surrounding epithelial lumen after one minute of IV exposure (2). Additionally, the same group reported being able to better characterize the vascularization of the tumor to further clarify the invasiveness of the cancer. ICG usage has been shown to be safe in a similar clinical setting by the Gotoh group, who used ICG to detect and characterize bullous and emphysematous lesion of the lung in video assisted thoracoscopic surgeries (VATS) with Infrared Thoracoscopy that were not previously detectable by white light (3).

The currently proposed trial is a single center, open-label pilot/observational cohort study. Patients with a diagnosis of resectable thoracic nodule/mass who are presumed to be resectable via minimally invasive surgery as determined by pre-operative assessment at the Hospital of the University of Pennsylvania will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age
2. Patients presenting with a thoracic nodule presumed to be resectable cancer on pre-operative assessment
3. Good minimally invasive operative candidates as determined by a thoracic oncology multidisciplinary team
4. Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

1. Pregnant women as determined by urinary or serum beta human chorionic gonadotropin (hCG) within 72 hours of surgery
2. Subjects with a history of iodide allergies
3. At-risk patient populations

   1. Homeless patients
   2. Patients with drug or alcohol dependence
   3. Children and neonates
   4. Patients unable to participate in the consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Ability of imaging system to detect expression of ICG in nodule/mass (i.e. tumor) and discern uptake of dye by tumor | 36 months
  Detected with imaging probe during minimally invasive procedure

SECONDARY OUTCOMES:
Incidence rates of all adverse events, treatment-emergent adverse events, and adverse device events from time of ICG administration through participants' first, post-operative appointment with surgeon | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Mountain CF, Dresler CM. Regional lymph node classification for lung cancer staging. Chest. 1997 Jun;111(6):1718-23. doi: 10.1378/chest.111.6.1718. PMID 9187199
- [Background] Kimura T, Muguruma N, Ito S, Okamura S, Imoto Y, Miyamoto H, Kaji M, Kudo E. Infrared fluorescence endoscopy for the diagnosis of superficial gastric tumors. Gastrointest Endosc. 2007 Jul;66(1):37-43. doi: 10.1016/j.gie.2007.01.009. PMID 17591472
- [Background] Gotoh M, Yamamoto Y, Igai H, Chang S, Huang C, Yokomise H. Clinical application of infrared thoracoscopy to detect bullous or emphysematous lesions of the lung. J Thorac Cardiovasc Surg. 2007 Dec;134(6):1498-501. doi: 10.1016/j.jtcvs.2007.07.051. PMID 18023672